CLINICAL TRIAL: NCT00460733
Title: Local (Brazil) Study, Multicenter, Opened, Comparative, Randomized, With Parallel Groups, Phase IV, in Post Menopausal Woman With Colles' Fracture of the Risedronate Sodium Usage in the Consolidation and in the Callus of the Colles'Fracture.
Brief Title: SOLID-Effect of Risedronate Sodium at Distal Radius in Colle's Fracture.
Acronym: SOLID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RISED_L_01930
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Colles' Fracture
MeSH Terms: conditions — Colles' Fracture | interventions — Risedronic Acid; Calcium

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Risedronate sodium
- 2 (Active Comparator)
  Interventions: Drug: Calcium & Vitamine D3

INTERVENTIONS:
Drug: Risedronate sodium — Actonel® 35 mg (risedronate sodium) and 1000 mg of calcium and 400 UI of Vitamine D3
  Arms: 1
Drug: Calcium & Vitamine D3 — 1000 mg of calcium and 400 UI of Vitamine D3
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of risedronate sodium (Actonel®) after a wrist fracture in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women with description of 2 or more years of Menopause;
* T-score <= -2.0 sd;
* Confirmed colles'fracture;
* Independent for the march (preserved ambulatorial ability);

Exclusion Criteria:

* Co-morbidities;
* Regular use of corticosteroids or other anti-resorptive drug in the last year;
* Use of drugs that can affect the calcium metabolism;
* Hypersensitivity to risedronate;
* Previous wrist or forearm fracture;
* Hypocalcemia;
* Renal insufficiency;
* Rheumatic disease;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2007-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Body mineral density of the 33% radius region and of the UD radius region | after 90 days of treatment

SECONDARY OUTCOMES:
Body mineral density of the 33% radius region and of the UD radius region | after 180 days of treatment
Size of callus obtained through Rx of the fracture site. | from the beginning up to the end of the study
Safety: Adverse events occurrence. | from the inform consent signature up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil